CLINICAL TRIAL: NCT05231954
Title: Digital Detection of Dementia (D Cubed) Studies: D2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, MALAZ BOUSTANI, Professor of Aging Research, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2008372812a; R01AG069765-01 (NIH)
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease and Related Dementias (ADRD)
MeSH Terms: conditions — Alzheimer Disease | interventions — Mass Screening; Patient Reported Outcome Measures

STUDY DESIGN:
Intervention Model Description: This is a pragmatic cluster randomized control trial with randomizing clinic and with wavier of consent for human subjects. The data collection is from the EHR. There is no research data collection outside the EHR.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Annual Well Visit or any other visit to Primary Care Doctor (No Intervention): Annual Well Visit or any other visit to Primary Care Doctor: This is the usual care arm. Electronic Health Record Data for patients from the clinics randomized to usual care will be collected for comparison with the other 2 arms. Patients from these primary care clinics must have had a visit to their doctor either as an annual well visit (AWV) or any other type of visit. These clinics will not have to do anything for the study but run their business as usual without altering anything.
- Passive Digital Marker (PDM) (Experimental): Passive Digital Marker (PDM): Electronic Health Record Data from those clinics randomized to PDM will be run through the PDM, a machine learning algorithm which can predict ADRD one year and three years prior to its onset.
  Interventions: Other: Passive Digital Marker for screening for ADRD
- Passive Digital Marker (PDM) + Quick Dementia Rating Scale (QDRS) (Active Comparator): Patients in the primary care clinics randomized to PDM+QDRS will have Electronic Health Record Data of their patients run through the PDM, a machine learning algorithm which can predict ADRD one year and three years prior to its onset. In addition, patients from these clinics will have their patients complete the QDRS, a validated patient reported outcome (PRO) tool. This combined approach will assess the value of early detection of ADRD and if the annual well visit can overcome the barriers related to early detection of ADRD.
  Interventions: Other: Passive Digital Marker for screening for ADRD

INTERVENTIONS:
Other: Passive Digital Marker for screening for ADRD — Patients in the primary care clinics randomized to PDM+QDRS will have Electronic Health Record Data of their patients run through the PDM, a machine learning algorithm which can predict ADRD one year and three years prior to its onset. In addition, patients from these clinics will have their patients complete the QDRS, a validated patient reported outcome (PRO) tool. This combined approach will assess the value of early detection of ADRD and if the annual well visit can overcome the barriers related to early detection of ADRD.
  Other Names: Patient reported outcome (QDRS) for screening for ADRD
  Arms: Passive Digital Marker (PDM); Passive Digital Marker (PDM) + Quick Dementia Rating Scale (QDRS)

SUMMARY:
The specific aim of the pragmatic trial is to evaluate the practical utility and effect of the PDM, the QDRS, and the combined approach (PDM + QDRS) in improving the annual rate of new documented ADRD diagnosis in primary care practices.

DETAILED DESCRIPTION:
Alzheimer's disease and related dementias (ADRD) negatively impact millions of Americans with an annual societal cost of more than $200 million.1 Currently, half of Americans living with ADRD never receive a diagnosis.2-7 For those who do, the diagnosis often occurs two to five years after the onset of symptoms.6-9 As stated by the National Institute on Aging (NIA) (RFA-AG-20-051) "The inability to diagnose and treat cognitive impairment results in prolonged and expensive medical care" and "early detection could help persons with dementia and their care partners plan for the future". Furthermore, if the development of disease modifying therapeutics for ADRD is successful, this may require the use of such therapeutics at a very early stage of ADRD.1 However, the current approaches of using cognitive tests or biomarkers for early detection of ADRD are not scalable due to their low acceptance, their invasive nature, their cost, or their lack of accessibility in rural or underserved areas. Thus, the NIA called out for the development of low cost, effective, and scalable approaches for early detection of ADRD (RFA-AG-20-051).

In response to the RFA-AG-20-051 call for the "validation, and translation of screening and assessment tools for measuring cognitive decline a pragmatic cluster-randomized controlled comparative effectiveness (NIH Stage IV) trial will be executed in Eskenazi Health in central Indiana and one additional replicated pragmatic trial among patients from diverse rural, suburban and urban primary care practices in south Florida. The pragmatic trial will incorporate the Passive Digital Marker (PDM) and the Quick Dementia Rating Scale (QDRS) within the Medicare paid Annual Wellness Visit (AWV) for a cohort of patients from practices across the two independent sites, with practices randomized in each pragmatic trial to one of the 3 arms (AWV alone, the AWV with PDM and the PDM and the QDRS).

Quick Dementia Rating Scale (QDRS)- is a validated patient reported outcome (PRO) tool.

Passive Digital Marker (PDM) - is a Machine Learning (ML) algorithm which can predict ADRD one year and three years prior to its onset by using routine care electronic health record (EHR) data. The algorithm was trained using structured and unstructured data from three EHR datasets: diagnosis (Dx), prescriptions (Rx), and medical notes (Nx). Individual algorithms derived from each of the three datasets were developed and compared to a combined one that included all three datasets.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* At least one visit to primary care practice within the past year
* Ability to provide informed consent
* Ability to communicate in English or Spanish
* Available EHR data from at least the past three years

Exclusion Criteria:

* Prior ADRD or mild cognitive impairment diagnosis as determined by ICD-10 code
* Evidence of any history of prescription for a cholinesterase inhibitors or memantine.
* Has serious mental illness such as bipolar or schizophrenia as determined by ICD-10 code
* Permanent resident of a nursing facility

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5325 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malaz Boustani, MD, MPH, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
We are collecting clinic based aggregated data.

REFERENCES:
- [Derived] Boustani MA, Ben Miled Z, Owora AH, Fowler NR, Dexter P, Puster E, Grout RW, Summanwar D, Erazo SF, Disla S, Coppedge K, Galvin JE. Digital Detection of Dementia in Primary Care: A Randomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2542222. doi: 10.1001/jamanetworkopen.2025.42222. PMID 41212562
- [Derived] Kleiman MJ, Plewes AD, Owora A, Grout RW, Dexter PR, Fowler NR, Galvin JE, Miled ZB, Boustani M. Digital detection of dementia (D3): a study protocol for a pragmatic cluster-randomized trial examining the application of patient-reported outcomes and passive clinical decision support systems. Trials. 2022 Oct 11;23(1):868. doi: 10.1186/s13063-022-06809-5. PMID 36221141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: D2 trial was launched at 9 clinics on July 5, 2022 (3 clinics in each study arm). D2 trial was completed in July 2024. The D2 trial deployed the Passive Digital Marker (PDM) on 5,325 older patients who were eligible and enrolled to receive primary care services within one of the 9 randomized clinics.
Pre-assignment Details: * At least 65 years old as of date of data pull.
  * At least 3 years of EHR data as of date of data pull.
  * Alive as of date of data pull.
  * No prior ADRD, MCI, bipolar, or schizophrenia diagnosis as determined by ICD-10 code.
  * No evidence for any history of cholinesterase inhibitors or memantine prescription."
  Within each clinic, enrolled patients include only those who:
  * Meet the above eligibility criteria
  * Have at least one visit to a randomized clinic during the study period.
Units Other Than Participants: Clinics
Period: Overall Study
Arm/Group | Annual Well Visit or Any Other Visit to Primary Care Doctor | Passive Digital Marker (PDM) | Passive Digital Marker (PDM) + Quick Dementia Rating Scale (QDRS)
Started | 1724; 3 Clinics | 1300; 3 Clinics | 2301; 3 Clinics
Completed | 1724; 3 Clinics | 1300; 3 Clinics | 2301; 3 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Population: * At least 65 years old as of date of data pull.
  * At least 3 years of EHR data available as of date of data pull.
  * Alive as of date of data pull.
  * No prior ADRD, MCI, bipolar, or schizophrenia diagnosis as determined by ICD-10 code.
  * No evidence for any history of cholinesterase inhibitors or memantine prescription."
  Enrolled patients include only those who:
  * Meet the above eligibility criteria
  * Have at least one visit to a randomized clinic during the study period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Annual Well Visit or Any Other Visit to Primary Care Doctor | Passive Digital Marker (PDM) | Passive Digital Marker (PDM) + Quick Dementia Rating Scale (QDRS) | Total
Number analyzed (Participants) | 1724 | 1300 | 2301 | 5325
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (6) | 71 (6) | 71 (6) | 71 (6)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex at birth.
  Participants
    Sex/Gender: Female | 1036 | 827 | 1449 | 3312
    Sex/Gender: Male | 688 | 473 | 852 | 2013
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 12 | 9 | 30
  Asian | 10 | 13 | 14 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 986 | 605 | 1336 | 2927
  White | 575 | 471 | 743 | 1789
  More than one race | 104 | 157 | 157 | 418
  Unknown or Not Reported | 40 | 42 | 42 | 124

OUTCOME MEASURES:

1. Primary Outcome: 12-Month Cumulative Incidence of ADRD Diagnoses
Description: Any new ADRD case identified (documented in the EHR) within 12 months of the Annual Wellness Visit (index visit).
Time Frame: 12 months after index visit
Population: 9 clinics were randomized, and patients were treated as per the randomization arm (3 clinics per arm)
Measure: Number; unit: Number of new ADRD cases
Arm/Group | Annual Well Visit or Any Other Visit to Primary Care Doctor | Passive Digital Marker (PDM) | Passive Digital Marker (PDM) + Quick Dementia Rating Scale (QDRS)
Number analyzed (Participants) | 1724 | 1300 | 2301
Number of new ADRD cases | 213 | 134 | 355
Statistical Analysis 1: Comparison: Annual Well Visit or Any Other Visit to Primary Care Doctor vs Passive Digital Marker (PDM) + Quick Dementia Rating Scale (QDRS); Test type: Superiority; p = 0.006, Mixed Models Analysis — P-value is adjusted for multiple comparisons, and a priori threshold for statistical significance is 0.05; Odds Ratio (OR) = 1.29, 95% CI 2-sided [1.08 to 1.55]
Statistical Analysis 2: Comparison: Annual Well Visit or Any Other Visit to Primary Care Doctor vs Passive Digital Marker (PDM); Test type: Superiority; p = 0.081, Mixed Models Analysis — The p-value is adjusted for multiple comparisons, and a priori threshold for statistical significance is 0.05; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.65 to 1.03]

2. Secondary Outcome: 12-Month Cumulative Incidence of ADRD Services
Description: The secondary outcome measures is receipt of any services related to cognitive diagnostic assessment in the post Annual Wellness Visit (index) period that providers may order to diagnose or exclude ADRD. Specifically, the metrics of diagnostic assessment are evaluated as proportions of patients with a record of 1 or more of:
  * Laboratory tests for TSH, serum B12, folate, or syphilis; individually or combined at any point during the 90 days after index
  * Neuropsychological testing, including testing by psychologist or physician, technician administrator, computer, or other providers during the 12 months after index date
  * Brain imaging testing (computed tomography, magnetic resonance imaging, positron emission tomography, magnetic resonance angiogram) of the head and neck, brain, or skull during the 12 months after index date
  * Medications approved for management of ADRD (cholinesterase inhibitors, memantine) during the 12 months after index date
Time Frame: 12 months after index visit
Population: 9 clinics were randomized, and patients were treated as per the randomization arm (3 clinics per arm)
Measure: Number; unit: Participants with ADRD related servicess
Arm/Group | Annual Well Visit or Any Other Visit to Primary Care Doctor | Passive Digital Marker (PDM) | Passive Digital Marker (PDM) + Quick Dementia Rating Scale (QDRS)
Number analyzed (Participants) | 1724 | 1300 | 2301
Participants with ADRD related servicess | 879 | 636 | 1366
Statistical Analysis 1: Comparison: Annual Well Visit or Any Other Visit to Primary Care Doctor vs Passive Digital Marker (PDM) + Quick Dementia Rating Scale (QDRS); Test type: Superiority; p = 0.044, Mixed Models Analysis — The p-value is adjusted for multiple comparisons, and the a priori threshold for statistical significance is 0.05; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.01 to 2.05]
Statistical Analysis 2: Comparison: Annual Well Visit or Any Other Visit to Primary Care Doctor vs Passive Digital Marker (PDM); Test type: Superiority; p = 0.919, Mixed Models Analysis — The p-value is adjusted for multiple comparisons and the a priori threshold for statistical significance is 0.05; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.69 to 1.50]

ADVERSE EVENTS:
Time Frame: 12-Months of follow-up after index visit (enrollment date)
Arm/Group | Annual Well Visit or Any Other Visit to Primary Care Doctor | Passive Digital Marker (PDM) | Passive Digital Marker (PDM) + Quick Dementia Rating Scale (QDRS)
All-Cause Mortality (participants affected / at risk) | 26/1724 | 7/1300 | 25/2301
Serious Adverse Events (participants affected / at risk) | 561/1724 | 398/1300 | 816/2301
Other Adverse Events (participants affected / at risk) | 0/1724 | 0/1300 | 0/2301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Annual Well Visit or Any Other Visit to Primary Care Doctor (N=1724) | Passive Digital Marker (PDM) (N=1300) | Passive Digital Marker (PDM) + Quick Dementia Rating Scale (QDRS) (N=2301)
Positive for PDM and had Hospitalization (General disorders) | 88/561 (88) | 65/398 (65) | 148/816 (148)
Positive for PDM and had ER visit (General disorders) | 243/561 (243) | 175/398 (175) | 392/816 (392)
Positive for PDM and had PCC visit (General disorders) | 561/561 (561) | 398/398 (398) | 816/816 (816)
Positive for PDM and had Memory clinic visit (General disorders) | 33/561 (33) | 33/398 (33) | 62/816 (62)
Positive for PDM and had NEW Dementia Diagnosis (General disorders) | 87/561 (87) | 70/398 (70) | 186/816 (186)
Positive for PDM and had NEW Depression Diagnosis (General disorders) | 31/561 (31) | 18/398 (18) | 32/816 (32)
Positive for PDM and had NEW Suicidal Ideation Diagnosis (General disorders) | 2/561 (2) | 1/398 (1) | 3/816 (3)
Positive for PDM and had NEW significant incapacity Diagnosis (General disorders) | 35/561 (35) | 29/398 (29) | 41/816 (41)

LIMITATIONS AND CAVEATS:
We had a delay in releasing the second cohort of the PDM by about 3 months due to enabling an HL7 process. This made it possible for Epic to run a program to flag PDM and PDM+QDRS automatically. For the first cohort, we manually entered the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT05231954/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT05231954/ICF_001.pdf